CLINICAL TRIAL: NCT03882515
Title: Evaluation Of Peripheral Muscle Oxygenation In Individuals With Muscular Idiopathic Pain Before And After Myofascial Release: A Randomized Controlled Trial
Brief Title: Evaluation Of Peripheral Muscle Oxygenation In Individuals With Muscular Idiopathic Pain With Myofascial Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Gilmar Moraes Santos, Clinical Professor, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Trapezium Spectroscopy
Record Dates: First submitted 2019-03-07; First posted 2019-03-20 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Trapezius Muscle Strain
Keywords: Neck Pain; Fascia; Modalities of Physiotherapy; Oxygenation
MeSH Terms: conditions — Neck Pain | interventions — Myofascial Release Therapy; Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Evaluation of peripheral muscle oxygenation in individuals with muscular idiopathic pain before and after myofascial release
  Interventions: Other: Myofascial Release
- Sham group (Sham Comparator): Evaluation of peripheral muscle oxygenation in individuals with muscular idiopathic pain before and after continuous surface slip technique
  Interventions: Other: Continuous Surface Slip Technique
- Control group (Active Comparator): Evaluation and reassessment of asymptomatic individuals
  Interventions: Other: Without intervention

INTERVENTIONS:
Other: Myofascial Release — With the right hand in hand exerts caudal pressure in the superior fibers of the muscle, both sides by a minute and a half each. In the ventral decubitus, apply pressure and slip from T12 to the base of the skull nine times. Thumb in the individual's acromion and with the other to hold the pressure and slide in the direction of the other acromion three times. Hand at the base of the skull and with the contralateral tenar region perform pressure and slip in caudal direction on both sides by three times. Hand at the base of the skull and with the contralateral thumb exerting pressure and slip of C3 the distal insertion of the upper fibers on both sides. Thumbs at the base of the skull, exerting lateral traction of the fascia in opposite directions. Dorsal decubitus, thumbs above clavicles, perform detachment of fibers for one and a half minutes. Patient sitting, support the head of the metacarpals beside the spinous process from T1 to T12 and exert pressure and slip three times each.
  Arms: Experimental group
Other: Continuous Surface Slip Technique — 1. Individual in the ventral decubitus, position the entire palmar surface bilaterally in the spinous process of T1 in the caudal direction, performing superficial smoothing in a smooth and rhythmic movement up to T12.
  2. Return of the hands from the caudal direction towards the cranial direction, bypassing the lateral borders of the trapezius muscle following the direction of the inferior, middle and superior fibers.
  3. Continue surface smoothing with a smooth and rhythmic movement until the distal insertion of the trapezius upper fibers into the skull and resume step 1 slowly and continuously for 10 minutes.
  Arms: Sham group
Other: Without intervention — Evaluation and re-evaluation without intervention
  Arms: Control group

SUMMARY:
Introduction: Neck Pain (NP) is considered a common idiopathic disorder in the general population. Oriented from incorrect executions during daily activities the DPO compromises the trapezius muscle that has a viscoelastic coating called fascia, which, in turn, is a soft tissue component, belonging to the connective tissue, that permeates the entire human body. During some activities that generate muscle overload, the fascia may undergo energy demands in which the local blood supply may be decreased, causing tissue hypoxia to result in pain. Decreased tissue blood supply could limit or prevent slippage of myofascial tissues. However, myofascial release can influence mechanoreceptors within the fascia, contributing to changes in local fluid dynamics, reducing excessive muscle tension, capillary constriction, and increasing local blood flow. One of the tools available for hemodynamic evaluation is the Near Infrared Spectroscopy (NIRS), which can quantify and capture variations in hemoglobin levels. Aim: To investigate whether myofascial release improves peripheral muscle oxygenation, pain intensity, and functional capacity of individuals with trapezius muscle pain. Methods: It is a clinical, parallel, randomized, double blind controlled trial with three groups that will be divided into: experimental, Sham and control. The instruments to be used in the research will be: Pressure Algometer, Neck Disability Index Questionnaire, Visual Analogue Scale (VAS), NIRS and Electromyograph. The experimental group will receive a myofascial release protocol for 20 minutes once weekly for six weeks. The Sham group will receive a continuous surface slip technique for the same time and frequency and the control will perform the evaluation and re-evaluation. Results: The present research is expected to increase peripheral muscle oxygenation, decrease pain threshold and improve quality of life after 6 weeks of intervention.

DETAILED DESCRIPTION:
This study will be a double-blind randomized controlled trial (evaluator and patient), parallel in three groups (experimental group, Sham and control). Participants will initially be evaluated by a trained investigator who will be blinded and assigned randomly (random numbers generated on the computer) block for the experimental, sham, and control groups by means of an opaque envelope draw. In group division, participants with pain may not be contemplated to participate in the myofascial release protocol intervention group. However, the research will count on a group that will be contemplated with the technique of continuous superficial sliding (massage), which in turn, the literature points out benefits and well-being in its application. Finally, a group of individuals without pain will be evaluated and reevaluated and evaluated as a means of preventing pain and reducing TM peripheral muscle oxygenation. When making the invitation to participate in the survey, individuals will not be required to participate if they do not agree, and therefore will not be penalized. Participants who agree to participate in the survey will sign a Free and Informed Consent Form (Annex I) and will be informed of the possibility of withdrawing from the survey at any stage, without penalty. The collection of the evaluation and intervention will be carried out in a salon Clinic School of Physiotherapy in the Center of Health and Sports Sciences (CEFID) of the State University of Santa Catarina (UDESC) in the city of Florianópolis - SC. All personal identification data of the participants will be preserved according to resolution of the national health council, taking into account the possibility of scientific dissemination of the results obtained. The risks of these procedures will be medium, since the participant may present muscle pain after the intervention protocol. To minimize these risks will be available, if necessary, attendance at the Clinic School of Physiotherapy. Volunteers of both sexes, aged from 18 years neck pain more specifically, in TM during daily or work activities. The sample will be selected in a non-probabilistic way for convenience, and the individuals will be divided into three groups: experimental, Sham and control. The control group will be formed by healthy individuals and will be paired with the experimental group according to age and gender taking into account that they are two relevant variables when addressing the fascia.

ELIGIBILITY:
Inclusion criteria:

The inclusion criteria for the two groups (experimental and Sham) in the research will be:

* Subjects of both sexes over 18 years of age;
* Subjects with pain in the trapezius muscle in the last three months without definite cause; Obs: They should present at least "moderate" pain in NDI sessions 1 and 3 in the subjective pain reported in VAS.

Exclusion Criteria:

The exclusion criteria for both groups will be:

* Neurological diseases;
* History of trauma or cervical spine surgeries;
* Clinical diagnosis of hernia or nerve compression;
* Previous physiotherapy (last three months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline deoxyhaemoglobin, oxyhaemoglobin and tissue oxygenation index at six weeks | Pre intervention and 6 weeks post intervention
  For the measurement of peripheral muscle oxygenation, near-infrared spectroscopy (PortaMon®, Artinis, The Netherlands) will be used. Near infrared spectroscopy depends primarily on two characteristics of human tissue. First, the relative transparency of the tissue to light and, secondly, the light absorption characteristics dependent on the oxygenation of hemoglobin. By using several different wavelengths, relative changes in hemoglobin concentration can be displayed continuously. It is a non-invasive, accessible, continuous measure, and can be performed in the laboratory, or even in the field and without the need of special infrastructure, since it has the portable format (ARTINIS MEDICAL SYSTEMS, 2017).

SECONDARY OUTCOMES:
Change from baseline normalized EMG at 6 weeks | Pre intervention, 3 weeks post intervention and 6 weeks post intervention
  The TeleMyo DTS Desk Receiver® (Noraxon USA Inc., Scottsdale, USA) electromyograph will be used for acquisition and processing of the electromyographic signals of the trapezius muscle with 16-bit resolution digital analogue converter and RRMC> 100 dB. The signals will be picked up at a sampling frequency of 2000 Hz, and stored by MR 3.2 software (Noraxon U.S.A. Inc., Scottsdale, USA). The electromyograph uses Direct Transmission System (DTS) technology, for surface EMG and other biomechanical sensors, which uses wireless technology for real-time data transmission. It has been used both to determine the time of onset of the muscular electrical activity as well as the intensity to which the muscle is active, that is, the amplitude of the activity (PERRY and BURNFIED, 1992).

OTHER OUTCOMES:
Change from baseline pain thresholds at 6 weeks | Pre intervention, 3 weeks post intervention and 6 weeks post intervention
  To evaluate pressure pain thresholds, a digital algometer (JTech Commander Algometer®, USA) will be used to allow the actual measurement of pain thresholds and tolerances. The Pressure Algometer features an easy-to-handle design (a visor and a tip) and fine resolution for clinical identification of changes in pain sensitivity. It provides an objective and efficient assessment for treatment planning and evolution monitoring (JTECH MEDICAL INDUSTRIES, 2017).
Change from baselien Neck Desability Index at 6 weeks | Pre intervention, 3 weeks post intervention and 6 weeks post intervention
  The Neck Desability Index is a ten-item questionnaire designed to assess functional disability and pain in the region of the cervical spine. The calculation of the scores is obtained by adding the points and then converting the result into value, considering only the items answered by the individual. For each section, the total possible score is 5: if the first statement is marked with the section score = 0, if the last statement is checked, 5. If all sections are marked the total score is calculated as follows: Example : 16 (total score) 50 (total score possible) x 100 = 32%. If a section is lost or not calculated: 16 (total score) 45 (total possible score) x 100 = 35.5%. Minimum Change Detectable (90% confidence): 5 points or 10% points.
Change from Visual Analog Scale at 6 weeks | Pre intervention, 3 weeks post intervention and 6 weeks post intervention
  One-dimensional instrument for the evaluation of the subjective intensity of pain. It is a line with the numbers numbered 0-10. At one end of the line is marked "no pain" and the other "worst pain imaginable" (MARTINEZ, et al., 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Gilmar M Santos, PhD, Principal Investigator — Santa Catarina State University
Locations (1):
- Santa Catarina State University, Florianópolis, Santa Catarina, Brazil

REFERENCES:
- [Derived] Dos Santos Amorim M, Sinhorim L, Baptistella do Nascimento I, Wagner J, de Paula Lemos F, Duarte Franca ME, Schleip R, Sonza A, Moraes Santos G. Peripheral muscle oxygenation, pain, and disability indices in individuals with and without nonspecific neck pain, before and after myofascial reorganization(R): A double-blind randomized controlled trial. PLoS One. 2024 Feb 9;19(2):e0292114. doi: 10.1371/journal.pone.0292114. eCollection 2024. PMID 38335169